CLINICAL TRIAL: NCT05315882
Title: Cytomegalovirus Infection, Indirect Effects and Mortality in Hematopoietic Stem Cell Transplantation With Cyclophosphamide Post-transplant
Brief Title: Cytomegalovirus Infection After HSCT and PT-CY as GVHD Prophylaxis >> GVHD PROPHYLAXIS ERA
Acronym: CY-CMV-2020
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: FIM-CIC-2020-01
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: CMV Infection
Keywords: CMV; PT-CY; allogeneic stem cell transplantation
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic stem cell transplantation: Observational, no interventional

SUMMARY:
Multicentre, observational, retrospective study to analyze the differences in CMVi pattern and recurrences between two groups of allogeneic HSCT patients (haplo vs no haplo HSCT), with intervention both postransplant cyclophosphamide as GvHD prophylaxis, using a database with information from historical clinic data.

DETAILED DESCRIPTION:
The overall aim of the study is to to analize CMVi after PTCy for GVHD prophylaxis, with a detailed description of CMVi and recurrences, direct and indirect consequences, in a HSCT population comparing two cohorts: haploidentical HSCT vs no haploidentical HSCT

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Period of HSCT: January 1st 2013 to December 31th 2018.
3. GvHD prophylaxis: Post-transplantation Cyclophosphamide (50 mg/Kg on days +3 and +4 or +3 and +5) and calcineurine inhibitors as GvHD prophylaxis.
4. Conditioning chemotherapy regimen and source of stem cells: myeloablative or reduced intensity TBF (Thiotepa 5 mg/Kg D -7-6, Fludarabine 50 mg/m2 D -5-4-3, Busulfan 3,2 mg/Kg D -4-3-2) starting on D-7 followed by peripheral blood or bone marrow infusion on day 0.

Exclusion Criteria:

1. Cord blood HSCT.
2. Antilymphocytic or anti thymocytic thymoglobulin as GvHD prophylaxis.
3. Alentuzumab as GvHD prophylaxis.

3. Sirolimus as GvHD prophylaxis.

4. HIV positive, HVC, HVB active or latent at HSCT.

5. CMV prophylaxis with letermovir.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 300 patients with hematological malignancies under HSCT from matched sibling donors, unrelated matched and mistmatched donor and haploidentical family donor using PT-CY and CNI as GVHD prophylaxis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence of CMVi in HSCT with PT-Cy and CMVi requiring pre-emptive therapy (significant CMVi) | 1 year
Median time to CMVi | 1 year
Cumulative incidence of PET-CMVi by day +100, +180 and +365. | 1 year
Overall survival by day +100, +180 and +365 | 1 year
Overall mortality by day +100, +180 and +365 | 1 year
Non-relapse mortality by day +100, +180 and +365 | 1 year

SECONDARY OUTCOMES:
CMV indirect effects incidence | 1 year
  Hospital admissions, secondary infections, secondary toxicity.
Incidence of CMVi recurrent episodes | 1 year
CMV disease | 1 year
CMV direct mortality | 1 year
Cumulative incidence of II-IV aGvHD | 1 year
Cumulative incidence of moderate-severe cGvHD | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MARIA JESUS PASCUAL, MD, Principal Investigator — HOSPITAL REGIONAL MALAGA / BMT UNIT
Locations (1):
- Maria Jesus Pascual, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
Communication at the EBMT 2022 Prague congress
Supporting Information: SAP, CSR
Time Frame: 19 March 2022
URL: https://www.ebmt.org/annual-meeting